CLINICAL TRIAL: NCT06940206
Title: Multidirectional Isometric Assessment of the Hip in Young Swimmers
Brief Title: Multidirectional Isometric Assessment of the Hip
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, Pablo Hernandez-Lucas, Associate professor in health sciences, University of Vigo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Cadera
Record Dates: First submitted 2025-04-13; First posted 2025-04-23 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Sports Physical Therapy; Hip; Assessment, Self

STUDY DESIGN:
Intervention Model Description: Validation of multidirectional isometric hip strength
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Validation of Isometric Assessment of the Hip in Swimmers (Other): Participants perform isometric tests (flexion, extension, ABD, ADD) to assess isometric hip strength at different basic movements over two sessions. Data is collected to evaluate the reliability and validity of these tests for swimmers.
  Interventions: Diagnostic Test: Multidirectional Isometric Assessment of the Hip

INTERVENTIONS:
Diagnostic Test: Multidirectional Isometric Assessment of the Hip — Participants perform isometric tests (flexion, extension, ABD, ADD) to assess isometric hip strength at different basic movements over two sessions. Data is collected to evaluate the reliability and validity of these tests for swimmers.

SUMMARY:
With the exception of the shoulder, the hip is among the most frequently injured areas in swimmers. Despite this, hip injuries are often overlooked in training and prevention programmes. Such neglect can cause significant damage to muscles, particularly the adductors, and the joint itself, potentially requiring arthroscopic surgery or even leading to secondary injuries in related structures such as the knee. Furthermore, hip strength and range of motion directly affect swimmers' underwater kicking speed. Although hip assessments are common in other sports, like football, for injury prevention and performance analysis-both dynamically and isometrically-isometric testing is particularly recommended due to its higher reproducibility.

Therefore, this study aims to validate a multidirectional isometric hip test in swimmers and examine agonist-antagonist muscle ratios in young advanced swimmers.

A comparative analysis will be conducted on 30 elite swimmers. This will include a descriptive analysis of the group and comparative analyses between breaststroke/non-breaststroke swimmers and between genders. Maximum isometric contractions of both lower limbs will be measured using a Chronojump force sensor (Boscosystem, Barcelona, Spain).

Athletes will stand on a step positioned centrally within a rack or cage, either laterally or frontally depending on the movement assessed (ABD-ADD or flexion-extension, respectively). They will grip the appropriate supports with their hands and perform three maximal efforts of each movement lasting 3 seconds, without compensatory actions (any attempt with compensations will be discounted). There will be a 20-second rest between attempts. All three attempts will be recorded.

To assess measurement reliability, tests will be repeated after 48 hours for subsequent comparison.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 14 and 18 years.
* Swimmers who train at least 15 hours weekly.
* Swimmers who have participated in the national championship this season.

Exclusion Criteria:

* Swimmers with any current hip or lower limb pathology.
* Swimmers who have required hip surgery.
* Swimmers who, for any other reason, are unable to complete an isometric maximal strength test.
* No ability to perform the Multidirectional Isometric Assessment of the Hip without compensatory movements.
* Refusal to sign informed consent (or legal guardian's consent for minors).

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-04-28 (Estimated); Primary Completion 2025-05-05 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Intraclass Correlation Coefficient (ICC) for Multidirectional Isometric Test. | Measured at two time points: baseline (Day 0) and follow-up (Day 2).
  Assessment of between-day reliability of the Multidirectional Isometric Test using intraclass correlation Coefficients (ICC) for hip flexion, extension, abduction and adduction movements.
Coefficient of Variation (CV) for Multidirectional Isometric Test. | Measured at two time points: baseline (Day 0) and follow-up (Day 2).
  Analysis of the coefficient of variation (CV) to evaluate data dispersion and consistency for Multidirectional Isometric Test.
Minimum Detectable Change (MDC) for Multidirectional Isometric Test. | Measured at two time points: baseline (Day 0) and follow-up (Day 2).
  Calculation of the minimum detectable change (MDC) to identify the smallest significant change in performance beyond measurement error for Multidirectional Isometric Test. (MDC90: Minimal Detectable Change at 90% Confidence; MDC%: Minimal Detectable Change Percentage).
Force Ratios Between for Multidirectional Isometric Test. | Measured at point baseline (Day 0).
  Evaluation of the agonist-antagonist strength ratios between hip flexion, extension, abduction and adduction movements.